CLINICAL TRIAL: NCT06893224
Title: Can the Belgian Coastal Environment Boost Physical and Cognitive Health in Older Adults?
Brief Title: Can the Belgian Coastal Environment Improve Physical and Cognitive Health in Older Adults?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0225
Record Dates: First submitted 2025-02-17; First posted 2025-03-25 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Physiologic Monitoring; Self-report Questionnaire; Sleep Quality; Cognitive Function
Keywords: Coastal environments; Older adults; Physiological stress; Cognitive function; Sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- First a coastal exposure followed by an urban exposure (Experimental): Participants assigned to this arm will first perform a coastal exposure (15 minutes of seated exposure, followed by 30 minute-walk), followed by an urban exposure a week later.
  Interventions: Other: Coastal exposure; Other: Urban exposure
- First an urban exposure, followed by a coastal exposure (Experimental): Participants assigned to this arm will first perform an urban exposure (15 minutes of seated exposure, followed by 30 minute-walk), followed by a coastal exposure a week later.
  Interventions: Other: Coastal exposure; Other: Urban exposure

INTERVENTIONS:
Other: Coastal exposure — This is a "real-life" exposure to the coastal environment, in which participants walk to a bench, sit there for 15 minutes, followed by a walk of approximately 30 minutes. After the 15 minute sitting period, a saliva sample is collected. During the walk, participants are equipped with wearable sensors. The walking route is indicated on a map.
Other: Urban exposure — This is a "real-life" exposure to the urban environment, in which participants walk to a bench, sit there for 15 minutes, followed by a walk of approximately 30 minutes. After the 15 minute sitting period, a saliva sample is collected. During the walk, participants are equipped with wearable sensors. The walking route is indicated on a map.

SUMMARY:
The goal of this interventional study is to learn if exposure to coastal environments improves the physical and cognitive health of older adults over the age of 60. The main questions it aims to answer are:

Does coastal exposure affect physical stress levels in older adults? Does coastal exposure affect self-reported stress levels in older adults? Does coastal exposure affect cognitive measures, such as sustained attention, in older adults? Does coastal exposure affect sleep quality in older adults? Is there a difference between the various components of coastal environments (e.g. dykes, dunes,...) in their effect on older adults' physical stress?

This wil be a within-subject study, in which participants get exposed to both a coastal and an urban environment to compare their response to these environments.

Participants will perform a coastal and urban walk on different days, equipped with wearable sensors (namely a wrist- and chestband) to measure various parameters such as heart rate and skin conductivity. Before, during and after the walk saliva samples will be collected for cortisol analysis. Before and after the walks they will also answer some questions (on e.g. overall demographics but also self-reported mental health) and perform cognitive tests (to study e.g. sustained attention).

DETAILED DESCRIPTION:
Due to practical reasons regarding time, infrastructure and resources, the second phase with video exposure was cancelled.

ELIGIBILITY:
Inclusion Criteria:

You are willing to make the time needed to complete the experiment. You understand and can communicate in Dutch. You are 60 years or older and retired. You are familiar with the city of Ostend. This means you visit Ostend multiple times per year and are preferably familiar with the area around the Grote Post and Fort Napoleon.

You smoke no more than 10 cigarettes per day. You are able and comfortable walking for approximately 30 minutes at an average pace without aids such as a cane or walker.

You do not have a pacemaker. You are not blind or deaf. You do not take tricyclic antidepressants or clozapine.

Exclusion Criteria:

People who cannot participate in the entire experiment, do not speak Dutch, are under 60 years old or not yet retired, have a pacemaker, are blind or deaf, take tricyclic antidepressants or clozapine, are not at all familiar with the city of Ostend, smoke more than 10 cigarettes per day, or are unable to walk for 30 minutes continuously without aids are not eligible to participate in the experiment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability - Time-domain measures | For a period of 2,5 to 3 hours
  During the entire protocol, both in the first and second phases of the study, interbeat intervals (IBIs) will be recorded using the Polar H10 chestband. From these IBIs, heart rate variability (HRV) measures will be calculated. Time-domain measures will be expressed in milliseconds (ms), including SDNN (Standard Deviation of NN intervals) and RMSSD (Root Mean Square of Successive Differences). These parameters provide insight into autonomic nervous system activity, particularly parasympathetic modulation.
Heart rate variability - Frequency-domain measures | For a period of 2,5 to 3 hours
  During the entire protocol, both in the first and second phases of the study, interbeat intervals (IBIs) will be recorded using the Polar H10 chestband. From these IBIs, heart rate variability (HRV) measures will be calculated. Frequency-domain measures, including low-frequency (LF) power, high-frequency (HF) power (expressed in milliseconds squared [ms²] or normalized units [nu]), and the LF/HF ratio (unitless), will be analyzed. These parameters provide insight into autonomic nervous system activity, with HF power primarily reflecting parasympathetic modulation and the LF/HF ratio indicating the balance between sympathetic and parasympathetic influences.
Electrodermal activity | For a period of 2,5 to 3 hours
  Electrodermal activity (EDA) of participants will be measured using the EmbracePlus wristband. EDA will be continuously recorded throughout the entire protocol, both during the first and second phases of the study. The primary EDA outcome measures include skin conductance level (SCL) and skin conductance responses (SCRs), both expressed in microsiemens (µS), These parameters provide insight into sympathetic nervous system activity and arousal dynamics.
Salivary cortisol | At 4 time points: before the exposure (baseline), after the seated exposure of 15 minutes, right after the walk, and 20 minutes after the walk
  Saliva samples will be collected in the first phase of the study, at 4 time points: before the exposure (baseline), after the seated exposure of 15 minutes, right after the walk, and 20 minutes after the walk. These saliva samples will be analysed for the presence of cortisol, which is expressed in nmol/L.
Sustained attention - Total number of items processed | Immediately before and immediately after the exposure to both environments (takes approximately 15 minutes)
  Sustained attention will be measured immediately before and after exposure to both environments, in both phases of the study. The validated d2 test of attention will be used for this. One outcome of this test is the total number of items processed (TN). This represents the total number of stimuli (letters) that a participant has scanned and attempted to process within the given time, with higher numbers indicating better sustained attention.
Sustained attention - Performance | Immediately before and immediately after the exposure to both environments (takes approximately 15 minutes)
  Sustained attention will be measured immediately before and after exposure to both environments, in both phases of the study. The validated d2 test of attention will be used for this. Another outcome of this test is the performance (P). This is calculated as the number of correctly marked target stimuli minus the number of errors (including both commission and omission errors). The higher this performance score, the better the participants' sustained attention.
Sustained attention - Error percentage | Immediately before and immediately after the exposure to both environments (takes approximately 15 minutes)
  Sustained attention will be measured immediately before and after exposure to both environments, in both phases of the study. The validated d2 test of attention will be used for this. Another outcome of this test is error percentage. This indicates the percentage of errors relative to the total number of marked items. Errors can be divided into: 1) commission errors (false positives) and 2) ommission errors (false negatives). Commision errors represent the incorrectly marked symbols that are not target stimuli. The ommission errors are the target stimuli that weren't marked. The lower the error percentage, the better participants' sustained attention.
Processing speed - Total correct responses | Immediately before and immediately after the exposure to both environments (takes approximately 15 minutes)
  Processing speed will be measured immediately before and after exposure to both environments, in both phases of the study. The validated Symbol Digit Modalities Test will be used for this. One outcome measure is the number of total correct responses. This is the number of correct symbol-digit pairings made within the given time limit. The higher this number, the better participants' processing speed.
Processing speed - Error rate | Before and after the exposure to both environments (takes approximately 15 minutes)
  Processing speed will be measured immediately before and after exposure to both environments, in both phases of the study. The validated Symbol Digit Modalities Test will be used for this. Another outcome measure of this test is the error rate, which is the number of incorrect responses. The lower the error rate, the better for participants' processing speed.

SECONDARY OUTCOMES:
Perceived stress | Immediately before and after exposure to both environments
  Perceived stress will be evaluated immediately before and after exposure to both environments. This will be measured using one question asking the participant "How stressed are you now?", which has to be scored on a ten-point Likert scale ranging from 1 (labelled "Not at all stressed") to 10 (labelled "Totally stressed").
Perceived mental exhaustion | Immediately before and after exposure to both environments
  Perceived mental exhaustion will be evaluated immediately before and after exposure to both environments. This will be measured using one question asking the participant "How mentally exhausted are you now?", which has to be scored on a ten-point Likert scale ranging from 1 (labelled "Not mentally exhausted at all") to 10 (labelled "Totally mentally exhausted").
Positive mood and negative mood | Immediately before and after exposure to both environments
  Positive mood will be evaluated immediately before and after exposure to both environments. This will be measured using the "Positive and Negative Affect Schedule". Participants will have to indicate to what extent they experience each of the emotions or feelings listed on a scale ranging from 1 (labelled "Very slightly or not at all") to 5 (labelled "Extremely").
Sleep quality | 14 days
  In the first phase of the study, participants will keep a sleeping diary for 14 days, to see whether the exposures to the different environments have an effect on their sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Mirko Petrovic, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No